CLINICAL TRIAL: NCT04110613
Title: A Randomized Controlled Trial to Reduce Periprocedural Fasting in Ventilated Trauma and Surgical Intensive Care Patients
Brief Title: RCT: Early Feeding After PEG Placement
Acronym: PEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Katie Love Bower, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-355
Record Dates: First submitted 2019-09-18; First posted 2019-10-01 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Critical Illness; Malnutrition; Gastrostomy; Procedural Sequelae; Trauma; Surgery; Mechanical Ventilation
MeSH Terms: conditions — Critical Illness; Malnutrition; Wounds and Injuries | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Once scheduled for the bedside PEG procedure, patients will be randomized to either the experimental NoFAST group or the control FAST group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- noFast: Start tube feeds within 1 hour of procedure (Active Comparator): The noFAST group will have post-PEG tube feeds initiated <1 hour after the procedure. Feeds are to be initiated at the rate and with the formula the patient was tolerating prior to the procedure.
  Interventions: Dietary Supplement: noFast: Start tube feeds within 1 hour of procedure
- FAST: Start tube feeds 4 hours after procedure (No Intervention): The FAST group will have post-PEG tube feeds initiated 4 hours after the procedure. Feeds are to be initiated at the rate and with the formula the patient was tolerating prior to the procedure.

INTERVENTIONS:
Dietary Supplement: noFast: Start tube feeds within 1 hour of procedure — Earliest possible initiation of tube feeding after bedside PEG tube procedure.
  Arms: noFast: Start tube feeds within 1 hour of procedure

SUMMARY:
Randomized controlled trial to establish evidence on which to base timing of enteral feeding after bedside PEG placement in ventilated Trauma and Surgical ICU patients.

DETAILED DESCRIPTION:
Trauma and surgical intensive care unit(TSICU) patients supported with mechanical ventilation are at high risk for complications associated with malnutrition (Ambrosino and Clini 2004; Aubier et al. 1985; Hill et al. 1998). To mitigate this risk, therapeutic enteral nutrition(EN) is delivered via nasogastric(NGT), orogastric(OGT), or nasoenteric tube(NET) as soon as possible after admission to the intensive care unit(ICU) or upon restoration of gastrointestinal(GI) continuity. Despite these interventions, TSICU patients often suffer a calorie deficit associated with enteral nutrition interruption(ENI) for procedures or transitions in care(Peev et al. 2015; McClave et al. 2009). These periods of fasting predict quantified caloric deficit associated with complications of malnutrition(Peev et al. 2015; Segaran, Barker, and Hartle 2016). Reduction in ENI duration before and after ICU procedures has yielded decreased caloric deficits within mixed ICU populations(Segaran, Barker, and Hartle 2016).

When the need for EN is prolonged, percutaneous endoscopic gastrostomy tube(PEG) placement is a bedside procedure employed to promote progress toward rehabilitation and disposition out of the ICU. First described in 1980, the technique found its success in replacing the classic open gastrostomy performed through a laparotomy incision under general anesthesia(Gauderer, Ponsky, and Izant 1980). Approximately 100,000-125,000 PEGs are performed annually in the United States(Mendiratta et al. 2012). Despite 40 years of experience and its routine nature in modern critical care settings, there is little evidence on which to base timing of tube feeds after PEG placement in the mechanically ventilated Trauma and Surgical ICU(TSICU) population.

Pre- and post-PEG tube placement fasting practices are highly variable among surgical intensivists. There is no standard of care, despite truncated periods of periprocedural fasting described as safe in previously published retrospective and prospective observational studies. There is no evidence to support prolonged fasting after PEG placement in TSICU patients, thus an opportunity to improve patient outcomes by providing evidence that will encourage earlier feeding and a reduction in calorie deficits.The aim of the study is to encourage a standard of care among surgical intensivists that will help to mitigate the risk of malnutrition in this highly susceptible patient population.

Trauma and Surgical ICU patients undergoing bedside PEG tube placement will be randomized to one of two groups: FAST and noFAST. The FAST group will have post-PEG tube feeds initiated 4 hours after the procedure. The noFAST group will have post-PEG tube feeds initiated <1 hour after the procedure. Feeds for both are to be initiated at the rate and with the formula the patient was tolerating prior to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over 18 years of age
* Negative pregnancy test for women participants of child-bearing age
* Mechanically ventilated surgical and trauma patients with clinical indication for PEG tube placement
* Tolerating tube feeds at goal prior to procedure

Exclusion Criteria:

* Patients with aberant gastrointestinal anatomy
* Patients with gastrointestinal motility disorders
* Patients with feeding intolerance prior to PEG tube procedure
* Pregnant women, children, or other vulnerable populations
* Clinical contraindications for PEG tube placement
* PEG performed in setting other than ICU at bedside

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hours fasted | 24 hours before to 72 hours after the procedure
  Number of hours patients are not receiving prescribed caloric intake

SECONDARY OUTCOMES:
Complications | 0-72 hours after the procedure
  Complications associated with timing to start tube feeds after bedside PEG placement
Calorie deficit | 24 hours to 72 hours after procedure
  Cumulative calorie deficit acquired as a result of peri-procedural fasting

CONTACTS AND LOCATIONS:
Overall Officials: Katie L Bower, MD, Principal Investigator — Carilion Clinic, Virginia Tech Carilion School of Medicine
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Peev MP, Yeh DD, Quraishi SA, Osler P, Chang Y, Gillis E, Albano CE, Darak S, Velmahos GC. Causes and consequences of interrupted enteral nutrition: a prospective observational study in critically ill surgical patients. JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):21-7. doi: 10.1177/0148607114526887. Epub 2014 Apr 7. PMID 24714361
- [Background] Segaran E, Barker I, Hartle A. Optimising enteral nutrition in critically ill patients by reducing fasting times. J Intensive Care Soc. 2016 Feb;17(1):38-43. doi: 10.1177/1751143715599410. Epub 2015 Feb 1. PMID 28979456
- [Background] Gauderer MW, Ponsky JL, Izant RJ Jr. Gastrostomy without laparotomy: a percutaneous endoscopic technique. J Pediatr Surg. 1980 Dec;15(6):872-5. doi: 10.1016/s0022-3468(80)80296-x. PMID 6780678
- [Background] Ali T, Le V, Sharma T, Vega KJ, Srinivasan N, Tierney WM, Rizvi S. Post-PEG feeding time: a web based national survey amongst gastroenterologists. Dig Liver Dis. 2011 Oct;43(10):768-71. doi: 10.1016/j.dld.2011.04.003. Epub 2011 May 31. PMID 21622036
- [Background] Stein J, Schulte-Bockholt A, Sabin M, Keymling M. A randomized prospective trial of immediate vs. next-day feeding after percutaneous endoscopic gastrostomy in intensive care patients. Intensive Care Med. 2002 Nov;28(11):1656-60. doi: 10.1007/s00134-002-1473-5. Epub 2002 Sep 6. PMID 12415457
- [Background] Gkolfakis P, Arvanitakis M, Despott EJ, Ballarin A, Beyna T, Boeykens K, Elbe P, Gisbertz I, Hoyois A, Mosteanu O, Sanders DS, Schmidt PT, Schneider SM, van Hooft JE. Endoscopic management of enteral tubes in adult patients - Part 2: Peri- and post-procedural management. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Feb;53(2):178-195. doi: 10.1055/a-1331-8080. Epub 2020 Dec 21. PMID 33348410
- [Background] Bechtold ML, Matteson ML, Choudhary A, Puli SR, Jiang PP, Roy PK. Early versus delayed feeding after placement of a percutaneous endoscopic gastrostomy: a meta-analysis. Am J Gastroenterol. 2008 Nov;103(11):2919-24. doi: 10.1111/j.1572-0241.2008.02108.x. Epub 2008 Aug 21. PMID 18721239
- [Background] Cobell WJ, Hinds AM, Nayani R, Akbar S, Lim RG, Theivanayagam S, Matteson-Kome ML, Choudhary A, Puli SR, Bechtold ML. Feeding after percutaneous endoscopic gastrostomy: experience of early versus delayed feeding. South Med J. 2014 May;107(5):308-11. doi: 10.1097/SMJ.0000000000000104. PMID 24937731
- [Background] Szary NM, Arif M, Matteson ML, Choudhary A, Puli SR, Bechtold ML. Enteral feeding within three hours after percutaneous endoscopic gastrostomy placement: a meta-analysis. J Clin Gastroenterol. 2011 Apr;45(4):e34-8. doi: 10.1097/MCG.0b013e3181eeb732. PMID 20733512
- [Background] Vyawahare MA, Shirodkar M, Gharat A, Patil P, Mehta S, Mohandas KM. A comparative observational study of early versus delayed feeding after percutaneous endoscopic gastrostomy. Indian J Gastroenterol. 2013 Nov;32(6):366-8. doi: 10.1007/s12664-013-0348-8. Epub 2013 Aug 17. PMID 23949988
- [Background] Dubagunta S, Still CD, Kumar A, Makhdoom Z, Inverso NA, Bross RJ, Komar MJ, Mulhisen L, Rogers JZ, Whitmire S, Whilden B. Early initiation of enteral feeding after percutaneous endoscopic gastrostomy tube placement. Nutr Clin Pract. 2002 Apr;17(2):123-5. doi: 10.1177/0115426502017002123. PMID 16214975
- [Background] Schneider AS, Schettler A, Markowski A, Luettig B, Kaufmann B, Klamt S, Lenzen H, Momma M, Seipt C, Lankisch T, Negm AA; *Conference presentation: 36th ESPEN Congress in Leipzig, Germany on August 31st - September 3rd, 2013. Complication and mortality rate after percutaneous endoscopic gastrostomy are low and indication-dependent. Scand J Gastroenterol. 2014 Jul;49(7):891-8. doi: 10.3109/00365521.2014.916343. Epub 2014 Jun 4. PMID 24896841
- [Background] Boullata JI, Carrera AL, Harvey L, Escuro AA, Hudson L, Mays A, McGinnis C, Wessel JJ, Bajpai S, Beebe ML, Kinn TJ, Klang MG, Lord L, Martin K, Pompeii-Wolfe C, Sullivan J, Wood A, Malone A, Guenter P; ASPEN Safe Practices for Enteral Nutrition Therapy Task Force, American Society for Parenteral and Enteral Nutrition. ASPEN Safe Practices for Enteral Nutrition Therapy [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jan;41(1):15-103. doi: 10.1177/0148607116673053. Epub 2016 Nov 5. PMID 27815525
- [Background] Blaser AR, Starkopf J, Kirsimagi U, Deane AM. Definition, prevalence, and outcome of feeding intolerance in intensive care: a systematic review and meta-analysis. Acta Anaesthesiol Scand. 2014 Sep;58(8):914-22. doi: 10.1111/aas.12302. Epub 2014 Mar 11. PMID 24611520
- [Background] ASGE Training Committee 2013-2014; Enestvedt BK, Jorgensen J, Sedlack RE, Coyle WJ, Obstein KL, Al-Haddad MA, Christie JA, Davila RE, Mullady DK, Kubiliun N, Kwon RS, Law R, Qureshi WA. Endoscopic approaches to enteral feeding and nutrition core curriculum. Gastrointest Endosc. 2014 Jul;80(1):34-41. doi: 10.1016/j.gie.2014.02.011. Epub 2014 Apr 26. No abstract available. PMID 24773773
- [Background] Ambrosino N, Clini E. Long-term mechanical ventilation and nutrition. Respir Med. 2004 May;98(5):413-20. doi: 10.1016/j.rmed.2003.11.008. PMID 15139570
- [Background] Aubier M, Murciano D, Lecocguic Y, Viires N, Jacquens Y, Squara P, Pariente R. Effect of hypophosphatemia on diaphragmatic contractility in patients with acute respiratory failure. N Engl J Med. 1985 Aug 15;313(7):420-4. doi: 10.1056/NEJM198508153130705. PMID 3860734
- [Background] Hill AT, Edenborough FP, Cayton RM, Stableforth DE. Long-term nasal intermittent positive pressure ventilation in patients with cystic fibrosis and hypercapnic respiratory failure (1991-1996). Respir Med. 1998 Mar;92(3):523-6. doi: 10.1016/s0954-6111(98)90302-x. PMID 9692116
- [Background] Sivasothy P, Smith IE, Shneerson JM. Mask intermittent positive pressure ventilation in chronic hypercapnic respiratory failure due to chronic obstructive pulmonary disease. Eur Respir J. 1998 Jan;11(1):34-40. doi: 10.1183/09031936.98.11010034. PMID 9543267